CLINICAL TRIAL: NCT06013904
Title: Can a Team of Ultrasound-Trained ED Physicians Reduce the Time to IV Placement for Children With Difficult IV Access?
Brief Title: Difficult PIV Placement in the Pediatric ED
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The logistics of the study made it too challenging to conduct within a pediatric setting.
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Lina Palomares, Project Manager, University of Texas at Austin
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 00004870
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual difficult PIV placement personnel (Active Comparator): Patients randomized to this arm will follow the usual protocol for difficult IV placement (ultrasound-trained nurses) in the pediatric ED.
  Interventions: Procedure: Difficult PIV placement personnel
- US-trained PEM Fellows (Experimental): Patients randomized to this arm will have a trained PEM fellow place the difficult PIV in the pediatric ED.
  Interventions: Procedure: US-trained PEM Fellows

INTERVENTIONS:
Procedure: Difficult PIV placement personnel — Patients randomized to this group will have their difficult PIV placed following the usual protocol for pediatric ED patients.
  Arms: Usual difficult PIV placement personnel
Procedure: US-trained PEM Fellows — US-trained PEM Fellows
  Arms: US-trained PEM Fellows

SUMMARY:
Insertion of peripheral intravenous (PIV) lines is one of the most common procedures in the Pediatric Emergency Department (ED). Faster placement of PIV lines can decrease time to intervention, as well overall time patients spend in the ED. Using ultrasound (US) guidance has been shown to increase the rate of first attempt success from around 50% to 78-85% compared to traditional methods of placing PIVs. The Pediatric ED at DCMC has US-trained nurses who assist in placing PIVs in patients with difficult access. Per ED shift, there is an average of 4-6 patients that are considered difficult access. However, because of nursing shortages and the general increased patient flow in the DCMC ED, there may not be a US-trained nurse available when a difficult access patient needs to have a PIV placed during a shift. This can lead to an increase in waiting time for the patient and delayed care.

At the DCMC ED, if the first attempt at placing a PIV is not successful, an algorithm for a level of escalation (i.e., which hospital personnel should attempt subsequent placements and maximum number of attempts) is followed. Attempt at PIV placement for most patients in the ED can be made by a patient care technician, RN, beside nurse, or charge nurse. If the PIV placement is not successful after two tries or if the patient has known risk factors that will complicate the PIV placement, the PIV placement is escalated to more experienced personnel, which includes US-trained nurses. For the purposes of this protocol, we will refer to these patients and personnel as Level 2 placements.

Pediatric emergency medicine (PEM) is a clinical subspecialty that focuses on caring for complicated and acutely ill pediatric patients in the emergency department. In partnership with Ascension Seton Dell Children's Medical Center, UT Austin's Dell Medical School PEM Fellowship is a rigorous program where Fellows are offered a broad experience in all facets of pediatric emergency medicine¸ including clinical care, teaching, research, and administration. A cohort of 12 Fellows are currently part of the program and could be trained to administer PIV via US, being available to place PIVs in patients with difficult access when a US-trained nurse is not available. We hypothesize that adding Pediatric Emergency Medicine (PEM) Fellows to the rotation of personnel who can insert IVs for pediatric patients with difficult access will shorten time to successful peripheral intravenous (PIV) placement overall in the Dell Children's Medical Center (DCMC) Emergency Department (ED).

ELIGIBILITY:
Inclusion Criteria:

1. Age 0-17
2. Patient meets difficult/escalated PIV criteria
3. English- or Spanish-speaking parent/guardian

Exclusion Criteria:

1. Critical illness presentation, such as sepsis.
2. Emergent medical situation, such as airway compromise, code, status epileptics, etc.

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Time to placement | During the patient 1 day visit, time to placement will be time from obtaining consent to successful IV placement saline flush.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Wilkinson, MD, MPH, Study Director — The University of Texas at Austin

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.